CLINICAL TRIAL: NCT05150756
Title: Intraoperative Lidocaine Infusion as a Sole Analgesic Versus Morphine in Laparoscopic Gastric Bypass Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada M.Samir, Assistant Professor of Anesthesia, Intensive care and Pain Management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R 35/ 2021
Record Dates: First submitted 2021-10-08; First posted 2021-12-09 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative
Keywords: lidocaine; morphine; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Lidocaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Lidocaine (Active Comparator): At induction of anesthesia, patients will receive a loading dose of intravenous (IV) 1.5mg/kg lidocaine hydrochloride 2% slowly over 3 min followed by IV infusion of 2mg/kg/hr lidocaine hydrochloride 2% via infusion pump. The infusion will be continued till the end of surgery.
  Interventions: Drug: Lidocaine Hydrochloride 2% Intravenous Solution [XYLOCAINE]
- Group Morphine (Active Comparator): At induction of anesthesia, patients will receive a loading dose of IV 0.1mg/kg morphine sulphate slowly over 3 minutes followed by IV infusion of normal saline via infusion pump. The infusion will be continued till the end of surgery
  Interventions: Drug: morphine sulphate (10mg/ ml ampoule)

INTERVENTIONS:
Drug: Lidocaine Hydrochloride 2% Intravenous Solution [XYLOCAINE] — At induction of anesthesia, patients will receive a loading dose of 1.5mg/kg lidocaine hydrochloride 2% slowly over 3 min followed by IV infusion of 2mg/kg/hr lidocaine hydrochloride 2% till the end of surgery
  Other Names: Xylocaine 2%
  Arms: Group Lidocaine
Drug: morphine sulphate (10mg/ ml ampoule) — At induction of anesthesia, patients will receive a loading dose of IV 0.1mg/kg morphine sulphate slowly over 3 minutes followed by IV infusion of normal saline via infusion pump. The infusion will be continued till the end of surgery
  Arms: Group Morphine

SUMMARY:
Postoperative opioid-centric pain management strategies in obese patients are accompanied by the possible development of; opioid-induced ventilatory impairment (OIVI) and hypoxemia. This presents as sedation and respiratory depression, combined with upper airway obstruction and hypercapnia. If it remains undetected and untreated, it can result in increased perioperative morbidity and mortality.Thus, an increased interest in the use of non-opioid analgesic adjuncts has been prompted.

Intra-operative intravenous lidocaine infusion has analgesic, anti-inflammatory, anti-hyperalgesic, opioid-sparing effects with an enhanced recovery after surgery (ERAS) profile. Its postoperative analgesia may last after reduction of its plasma concentration. So, lidocaine could be a good alternative in bariatric surgery.

Lidocaine has been studied as part of an opioid-free multimodal analgesia in morbidly obese patients. Also, its use in bariatric surgery showed a decrease in postoperative opioid use and improvement in the quality of recovery.

DETAILED DESCRIPTION:
compare the postoperative analgesic effect of intraoperative lidocaine infusion (Study group) used as a sole analgesic agent, to the intraoperative intravenous morphine (Control group) in laparoscopic gastric bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I- II
* body mass index (BMI) ˃ 35
* scheduled to undergo laparoscopic gastric bypass

Exclusion Criteria:

* Patients' refusal
* hypersensitivity to the study medications
* patients with known history of; hepatic disease, renal dysfunction
* severe renal impairment (eGFR <30ml/min/1.73m2)
* heart failure; left ventricular ejection fraction than 35%
* any cardiac dysrhythmias; Adam-Stokes syndrome; Wolff- Parkinson-White syndrome, atrio-ventricular block with heart rate below 50 bpm
* chronic pain
* concomitantly taking beta blocking drugs •substance abuse disorder
* chronic opioid use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Post-operative pain score at rest | 1hour
  Intensity of pain will be monitored ; on arrival to the PACU, at 20, 40 and 60 minutes after arrival to the PACU by the Numeric Pain Rating Scale. The Numeric Pain Rating Scale (NPRS) is a segmented numeric version of the visual analog scale (VAS) in which the patient selects a whole number (0-10 integers) that best reflects the intensity of pain felt.Where 0 is no pain felt and 10 is the worst pain.

SECONDARY OUTCOMES:
Duration of surgery | 3 hours
  measured in minutes
Duration of anesthesia | 4 hours
  measured in minutes
mean values of mean blood pressure (MBP) | 5 hours
  mean values of MBP will be recorded as base line value, before induction of anesthesia, 5 minutes after endotracheal intubation, before pneumoperitoneum, after release of pneumoperitoneum and 10 min after extubation in the PACU
Number of patients requiring intra-operative morphine | 4hours
  Number of patients requiring intra-operative morphine will be recorded
sPO2 | 5 hours
  recorded in the induction room and in the PACU.
Respiratory rate | 5 hours
  recorded in the induction room and in the PACU
Post-operative nausea and/or vomiting | 1 hour
  number of patients will be recorded
Post-operative sedation score | 1 hour
  From 0 to 4
Modified Aldrete Score | 1 hour
  score from 0 to 10. Higher score means patient is fit to transfer to the ward. In the PACU, patients with score ≥ 9 will be transferred to the surgical unit
mean values of heart rate (HR) | 5 hours
  mean values of HR will be recorded as base line value, before induction of anesthesia, 5 minutes after endotracheal intubation, before pneumoperitoneum, after release of pneumoperitoneum and 10 min after extubation in the PACU
Number of patients requiring postoperative additional morphine doses | 1 hour
  Number of patients requiring postoperative additional morphine doses willbe recorded
the total dose of morphine given to each patient | 5 hours
  the total dose of morphine given to each patient will be recorded in milligrams

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No